CLINICAL TRIAL: NCT02519686
Title: The Impact of Trendelenberg Positioning as Compared to Left Lateral Positioning on Ease of Colonoscope Insertion During Colonoscopy
Brief Title: Trendelenberg Versus Left Lateral Position for Colonoscopy
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201504136
Record Dates: First submitted 2015-07-13; First posted 2015-08-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Trendelenburg position maneuver: Trendelenburg (TD) positioning (supine with head tilt-down) is used in abdominal and gynecological surgery as well as during colonoscopy to allow better access to the pelvic organs, as gravity pulls the bowel out of the pelvic cavity and the rectosigmoid angle straightens.
- Left lateral position maneuver: Left Lateral (LL) position (patient laying on their side, traditionally used for colonoscopies)

SUMMARY:
The purpose of this study is to determine if the trendelenberg (TD) position (position in procedures that involves placing the patient at an angle so that their head is lower than their feet on the procedure bed) in select patients undergoing colonoscopy is superior than the left lateral (LL) position (patient laying on their side, traditionally used for colonoscopies) in terms of decreasing time necessary to pass the colonoscope through the left colon, and decreasing the difficulty of the procedure.

DETAILED DESCRIPTION:
The colonoscopists will be asked to rate their prediction of difficulty of the procedure prior to the colonoscopy and to rate the ease of procedure after the colonoscopy. The clinical experience of the study investigators is that TD positioning is superior to LL positioning in patients with risk factors for having a difficult colonoscopy (thin women; those with diverticulosis- small bulging pouches present in the colon; or prior pelvic surgery).

Patients with risk factors for difficult colonoscopy will be randomized to undergo colonoscopy while positioned in the TD position or the LL position during advancement of the colonoscope through the sigmoid colon. The sigmoid colon is a section of the colon, proximal to the rectum, that is curved. The sigmoid colon is a normal component of GI tract anatomy, although due to it's shape, especially with the risk factors listed previously; can cause challenges to inserting the colonoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Personal history of pelvic surgery
2. Diverticulosis, identified by patient report or review of previous colonoscopy or imaging studies.
3. BMI < 25.

Exclusion Criteria:

1. Patients who do not meet inclusion criteria.
2. Patients who have undergone colonic resection
3. Patients with glaucoma
4. Patients with uncontrolled acid reflux disease or active nausea/vomiting.
5. Patients who are unwilling or unable to consent.
6. BMI > 30

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cecal insertion time | intraoperaive
  The time from scope insertion to the cecum

CONTACTS AND LOCATIONS:
Overall Officials: Dayna S Early, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Thorlakson RH, Thorlakson TK. The lithotomy-Trendelenburg position for restorative resection by stapling and abdominoperineal excision of the rectum. Can J Surg. 1984 May;27(3):246-7. PMID 6372977
- [Background] Ozcan MS, Praetel C, Bhatti MT, Gravenstein N, Mahla ME, Seubert CN. The effect of body inclination during prone positioning on intraocular pressure in awake volunteers: a comparison of two operating tables. Anesth Analg. 2004 Oct;99(4):1152-1158. doi: 10.1213/01.ANE.0000130851.37039.50. PMID 15385367
- [Background] Shah HA, Paszat LF, Saskin R, Stukel TA, Rabeneck L. Factors associated with incomplete colonoscopy: a population-based study. Gastroenterology. 2007 Jun;132(7):2297-303. doi: 10.1053/j.gastro.2007.03.032. Epub 2007 Mar 21. PMID 17570204
- [Background] Weinstock LB, Early DS. Colonoscopy in the tilt-down position. Gastrointest Endosc. 2014 Oct;80(4):746. doi: 10.1016/j.gie.2014.05.328. No abstract available. PMID 25220519